CLINICAL TRIAL: NCT02063542
Title: Cerebrospinal Fluid Cholinergic Biomarkers and Postoperative Cognitive Change in Aged Patients
Brief Title: CSF Cholinergic Biomarkers and Postoperative Cognitive Change
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, diansan su, Principal Investigator, RenJi Hospital
Other Study IDs: ACHandPOCD
Record Dates: First submitted 2014-02-08; First posted 2014-02-14 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Necrosis of Femoral Head; Knee Osteoarthritis; Fracture of Lower Limb
Keywords: Postoperative cognitive changes; Acetylcholine in CSF; Surgery
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebral spinal fluid
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Previous study demonstrated that the condition of central cholinergic nerve is important for the postoperative cognitive dysfunction. In present study investigators hypothesized that the acetylcholine concentration in the cerebral spinal fluid is associated to the postoperative cognitive changes in aged patients undergoing osteopathic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elder than 60 years old
* Spoke proficient Mandarin Chinese
* Agree to undergoing spinal plus general anesthesia
* Selected total knee replacement surgery

Exclusion Criteria:

* Patients with neurological and/or psychiatric diseases, including AD, stroke and psychosis
* Have contraindication for spinal anesthesia such as clotting disorder local infection in the puncture site
* Existing cognitive impairment as evidenced by Mini-Mental State Examination scores below 24
* Several audition or vision disorder
* Unwillingness to comply with the protocol or procedures.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aged patients undergoing total knee replacement surgery.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Short-term postoperative cognitive dysfunction rate | The day before surgery and 7 days after surgery (or before leave hospital)
Concentration of Acetylcholine in CSF | During spinal anesthesia
Concentration of choline acetyltransferase in CSF | During spinal anesthesia
Concentration of acetylcholinesterase in CSF | During spinal anesthesia

SECONDARY OUTCOMES:
Long-term postoperative cognitive dysfunction rate | Two months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Dr., Study Chair — Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China